CLINICAL TRIAL: NCT07101965
Title: Phase I Clinical Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RSS0343 Tablets in Healthy Subjects After Single and Multiple Oral Administration and the Effect of Food on the Pharmacokinetics of RSS0343
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSD51318
Record Dates: First submitted 2025-07-13; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Health Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Treatment group 1: RSS0343 tablets or placebo (Experimental)
  Interventions: Drug: RSS0343 tablets ；placebo
- Treatment group 2: RSS0343 tablets or placebo (Experimental)
  Interventions: Drug: RSS0343 tablets ；placebo
- Treatment group 3: RSS0343 tablets or placebo (Experimental)
  Interventions: Drug: RSS0343 tablets ；placebo
- Treatment group 4: RSS0343 tablets or placebo (Experimental)
  Interventions: Drug: RSS0343 tablets ；placebo
- Treatment group 5: RSS0343 tablets or placebo (Experimental)
  Interventions: Drug: RSS0343 tablets ；placebo
- Treatment group 6: RSS0343 tablets or placebo (Experimental)
  Interventions: Drug: RSS0343 tablets ；placebo
- Treatment group 7: RSS0343 tablets or placebo (Experimental)
  Interventions: Drug: RSS0343 tablets ；placebo
- Treatment group 8: RSS0343 tablets or placebo (Experimental)
  Interventions: Drug: RSS0343 tablets ；placebo

INTERVENTIONS:
Drug: RSS0343 tablets ；placebo — RSS0343 tablets and placebo were given orally as a single dose
  Arms: Treatment group 1: RSS0343 tablets or placebo; Treatment group 2: RSS0343 tablets or placebo; Treatment group 3: RSS0343 tablets or placebo; Treatment group 4: RSS0343 tablets or placebo; Treatment group 5: RSS0343 tablets or placebo
Drug: RSS0343 tablets ；placebo — RSS0343 tablets and placebo were taken orally multiple times
  Arms: Treatment group 6: RSS0343 tablets or placebo; Treatment group 7: RSS0343 tablets or placebo; Treatment group 8: RSS0343 tablets or placebo

SUMMARY:
To evaluate the safety and tolerability of RSS0343 tablets in healthy subjects after single and multiple oral administration

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-55 years old (inclusive), male or female;
2. Body mass index in the range of 19-28 kg/m2 (inclusive).

Exclusion Criteria:

1. The results of physical examination, vital signs, laboratory tests, chest imaging, abdominal B ultrasound and 12-lead electrocardiogram were abnormal.
2. Hepatitis B surface antigen, hepatitis C antibody, syphilis antibody, HIV antibody positive;
3. Suspected allergy to the study drug or any component of the study drug, or severe allergy to any drug, food, toxin or other exposure;
4. Current active, latent, or inadequately treated M. tuberculosis (i.e., tuberculosis [TB]) infection;
5. Investigator-assessed clinically significant infection (e.g., requiring hospitalization or parenteral antimicrobial therapy) within 1 month before screening; A history of more than one previous episode of herpes zoster, or disseminated herpes zoster (one episode); Any history of other infections that the investigator considered might have been aggravated by study participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-04-07 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
adverse events | The observation lasted until the 61th day

SECONDARY OUTCOMES:
Cmax | The observation lasted until the 33th day
AUC0-t | The observation lasted until the 33th day
AUC0-inf | The observation lasted until the 33th day
Tmax | The observation lasted until the 33th day
t1/2 | The observation lasted until the 33th day
CL/F | The observation lasted until the 33th day
Vz/F | The observation lasted until the 33th day
Ae,urine | The observation lasted until the 33th day
fe,urine | The observation lasted until the 33th day
Relative bioavailability of premeal and postmeal administration | The observation lasted until the 16th day
Neutrophil elastase (NE) activity in peripheral blood after repeated oral administration of RSS0343 | The observation lasted until the 61th day

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital), Shandong, Jinan, China

IPD SHARING:
Plan to Share IPD: Undecided